CLINICAL TRIAL: NCT01010178
Title: Combination of Approved Drug in COPD
Brief Title: Can Airflow Limitation in Chronic Obstructive Pulmonary Disease (COPD) be Reversible by Drugs?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Responsible Party: Corresponding Author: Research Center of Chemical Injuries, Baqiyatallah Medical Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: BMT-1388-2
Record Dates: First submitted 2009-11-06; First posted 2009-11-09 (Estimated); Last update posted 2009-11-09 (Estimated); Status verified 2009-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Macrolid; reversibility; Theophylline; Corticosteroids; symptoms PFT
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Theophylline

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Macrolid, Theophylline, Corticosteroids (Experimental): Approved drug in this setting
  Interventions: Drug: Macrolid, Theophylline, Inhaler Corticosteroids

INTERVENTIONS:
Drug: Macrolid, Theophylline, Inhaler Corticosteroids — we have no permission to include them in detail because of privacy policy of mentioned journal for publication

SUMMARY:
Critical combination of various approved drugs in management for patients suffering with COPD.

ELIGIBILITY:
Inclusion Criteria:

* current or past smoker COPD

Exclusion Criteria:

* history of significant occupational or other environmental exposures or a connective tissue disease

Ages: 22 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2008-02; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
15% increasing in forced expiratory volume in 1 second | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Research Center of Chemical Injuries, Baqiyatallah Medical Sciences University, Mollasadra St,, Tehran, Iran